CLINICAL TRIAL: NCT04253145
Title: Phase I-II Study to Assess the Safety, Tolerability and Efficacy of PM01183 and Atezolizumab in Patients With Advanced Small Cell Lung Cancer That Progressed Following Prior Therapy With Platinum-Based Chemotherapy.
Brief Title: Study to Assess Safety,Tolerability,Efficacy of PM01183 and Atezolizumab in Patients w/ Advanced Small Cell Lung Cancer.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Oncosur (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2SMALL
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Small Cell Lung
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183; atezolizumab

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, uncontrolled and multicenter phase I-II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM01183 w/ Atezolizumab (Experimental): Patients will receive atezolizumab at a fixed dose of 1200 mg intravenously (i.v.) as a 60-minute infusion (the second and subsequent infusions may be administered over 30 minutes) followed by PM01183 at a starting dose of 2.5 mg/m2 i.v. as a 1-hour infusion on Day 1 every three weeks (q3wk). Following analysis of cohorts, dose levels can be escalated from 2.5mg to 3.2, to a maximum dose of 3.5 mg of PM01183
  Interventions: Drug: PM 01183; Drug: Atezolizumab

INTERVENTIONS:
Drug: PM 01183 — Lyophilisate for solution for infusion
  Other Names: Lurbinectidin
Drug: Atezolizumab — Concentrate for solution for infusion
  Other Names: Tecentriq

SUMMARY:
Prospective, open-label, uncontrolled and multicenter phase I-II study in SCLC patients with ECOG PS 0-1 who have failed one prior platinum-containing line but no more than one chemotherapy-containing line. The study will be divided into two parts: a dose-ranging phase I with escalating doses of PM01183 in combination with a fixed dose of atezolizumab, followed by a single-arm phase II part with expansion at the RD determined during the phase I.

DETAILED DESCRIPTION:
Phase I Patients will receive atezolizumab at a fixed dose of 1200 mg intravenously (i.v.) followed by PM01183 at a starting dose of 2.5 mg/m2 i.v. as a 1-hour infusion on Day 1 every three weeks (q3wk). PM01183 doses will be escalated in successive cohorts of patients following a modified Fibonacci scheme and a classical 3+3 design, and according to observed tolerance and safety.

Phase II Patients will receive atezolizumab i.v. as a 60-minute infusion (the second and subsequent infusions may be administered over 30 minutes) followed by PM01183 i.v. as a 1-hour infusion on Day 1 q3wk, at the RD determined during the phase I part.

It is expected that approximately 50% of patients included were previously treated with chemotherapy and the other 50% with immunotherapy and chemotherapy. In case one of the groups reaches 50% of the total number of patients expected to be recruited, no further patient will be included in this group and accrual will be limited to patients with the other group.

It is expected that approximately 50% of the patients included in the phase II part will be platinum-resistant [i.e., chemotherapy-free interval (CTFI) 30 to < 90 days from the end of first-line platinum-based chemotherapy] and 50% will be platinum-sensitive (i.e., CTFI ≥ 90 days), so as to assess efficacy in both settings. However in case that one of the CTFI groups reaches 60% of the total number of patients expected to be recruited, no further patient will be included in this group and accrual will be limited to patients with the other CTFI group.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated written informed consent prior to any specific study procedure.
* Age >18 years.
* Histologically or cytologically confirmed diagnosis of extensive or limited SCLC.
* Progression to first-line platinum-based chemotherapy. For phase II part: Progression to first- line platinum-based chemotherapy or first- line platinum- based chemotherapy and immunoterapy (anti PD1/ PDL1). A chemotherapy and/ or immunotherapy- free interval (CTFI, time from the last dose of first-line chemotherapy to the occurrence of progressive disease) ≥ 30 days.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score ≤1.
* Measurable disease according to RECIST v.1.1. Note: irradiated lesions may qualify as target if progression has been documented.
* At least three weeks since last prior anticancer treatment (including radiotherapy) and recovery to grade ≤ 1 from any adverse event (AE) related to previous anticancer treatment (excluding sensory neuropathy, anemia, asthenia and alopecia, all grade ≤ 2) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, v.5).
* Adequate bone marrow, renal, hepatic, and metabolic function (assessed ≤7 days before inclusion in the study):
* Platelet count ≥100 x 109/L, hemoglobin ≥9.0 g/dL and absolute neutrophil count (ANC) ≥1.5 x 109/L.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 x the upper limit of normal (ULN), independently of the presence of liver metastases.
* Alkaline phosphatase (AP) ≤2.5 x ULN.
* Total bilirubin ≤1.5 x ULN or direct bilirubin ≤ULN
* International Normalized Ratio (INR) <1.5 (except if patient is on oral anticoagulation therapy).
* Calculated creatinine clearance (CrCL) ≥30 mL/minute (using Cockcroft and Gault´s formula).
* Creatine phosphokinase (CPK) ≤2.5 x ULN.
* Albumin ≥3.0 g/dL. Albumin infusion to fulfill the inclusion criterion is forbidden.
* Thyroid stimulating hormone (TSH) within institutional normal limits. If TSH is above the ULN, then a free T4 within institutional normal limits is acceptable.
* Evidence of non-childbearing status for women of childbearing potential (WOCBP). Both women and men must agree to use a highly effective contraceptive measure during the trial, for at least five months after last atezolizumab dose, and for at least six weeks (women) or 4 months (men) after last PM01183 dose. Fertile male patients with WOCBP partners must agree to refrain from fathering a child or donating sperm during the trial and up to five months after treatment discontinuation. Acceptable methods of contraception include abstinence, intrauterine device (IUD), oral contraceptive, subdermal implant and/or double barrier.

Exclusion Criteria:

1. Active or untreated central nervous system (CNS) involvement. Treated CNS metastases have to show radiographic stability (defined as no CNS progression for at least three weeks from post-radiotherapy brain scan to brain scan performed prior study entry), and patients should not have neurologic sign/symptoms secondary to the brain metastases or RT. Any steroid treatment must be completed ≥ 14 days before first dose of study treatment.
2. More than one prior chemotherapy-containing line (re-challenge with the same initial regimen is not allowed).
3. Patients with radiation therapy (RT) in more than 35% of the bone marrow.
4. History of previous bone marrow and/or stem cell transplantation.
5. Impending need for RT (e.g., painful bone metastasis and/or risk of spinal cord compression).
6. History of allergy or hypersensitivity to any of the study drugs or their excipients.
7. Prior therapy with PM01183, antibodies against PD-1, PD-L1, PD-L2, CD137, or cytotoxic T lymphocyte associated antigen-4 (CTLA-4). For phase II part: Prior therapy with PM01183, PD-L2, CD137, or cytotoxic T lymphocyte associated antigen-4 (CTLA-4).
8. Live vaccines within 30 days prior to start of study treatment and while on treatment.
9. History of other prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer. Patients with other prior malignancies and no disease recurrence for 3 years are eligible.
10. Concomitant diseases/conditions:

    1. History or presence of unstable angina, myocardial infarction, congestive heart failure defined as abnormal left ventricular ejection fraction (LVEF) < 50% assessed by multiple-gated acquisition scan (MUGA) or equivalent by ultrasound (US), or clinically significant valvular heart disease within 12 months prior first study dose.
    2. Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment.
    3. Ongoing chronic alcohol consumption, or cirrhosis with Child-Pugh score B or C.
    4. Active uncontrolled infection. Serious non-healing wound, ulcer or bone fracture.
    5. Diagnose of immunodeficiency or receiving systemic steroids therapy (more than a daily dose of 10 mg of prednisone or equivalent per day) or any other form of immunosuppressive therapy within 14 days prior to the first study dose.
    6. Active autoimmune disease that required systemic treatment in the past two years (i.e., with disease-modifying agents, corticosteroids and immunosuppressive drugs).

       Patients with vitiligo or resolved childhood asthma/atopy are eligible, as well as patients who require intermittent use of bronchodilators or local steroid injections, patients with hypothyroidism stable on hormone replacement, patients with insulin-treated controlled type 1 diabetes or Sjogren's syndrome.
    7. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis or evidence of active pneumonitis on screening chest computed tomography (CT) scans. A history of radiation pneumonitis in radiation field (fibrosis) will be allowed if asymptomatic and not requiring steroids.
    8. Known history of active tuberculosis (Mycobacterium tuberculosis).
    9. Ongoing treatment-requiring, non-neoplastic chronic liver disease of any origin. For hepatitis B, this includes positive tests for both Hepatitis B surface antigen (HBsAg) and quantitative Hepatitis B polymerase chain reaction (PCR). For hepatitis C, this includes positive tests for both Hepatitis C antibody and quantitative Hepatitis C PCR. Patients taking hepatitis-related antiviral therapy within 6 months prior to the first study dose will also be excluded.
    10. Known human immunodeficiency virus (HIV) infection.
    11. Myopathy or any clinical situation that causes significant and persistent elevation of CPK (>2.5 x ULN in two different determinations performed one week apart).
    12. Limitation of the patient's ability to comply with the treatment or follow-up procedures.
    13. Patiens who have previously experienced pericarditis, pericardial effusion and cardiac tamponade) on prior treatment with other immune- stimulatory anticancer agents.
    14. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
11. Active COVID19 infection determined by PCR (positive result of SARS-CoV-2 virus), not mandatory if fully vaccinated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Determination of Maximum Tolerable Dose | one cycle - 21 days
  The MTD will be the lowest dose level explored during dose escalation at which more than one third of evaluable patients experience a DLT during Cycle 1.
Determination Recomended Dose: | one cycle - 21 days
  The RD will be the highest dose level explored during dose escalation at which less than one third of evaluable patients experience a DLT during Cycle 1.

SECONDARY OUTCOMES:
Progression-free survival | the time from the date of registration to the date of documented progression per RECIST v.1.1 or death, assessed approximately up to 30 months
  the time from the date of registration to the date of documented progression per RECIST v.1.1 or death. If the patient receives further antitumor therapy or is lost to follow-up before PD, PFS will be censored at the date of last tumor assessment before the date of subsequent antitumor therapy.
Duration of response | from the date of first documentation of response per RECIST v.1.1 (complete or partial response, whichever comes first) to the date of documented PD or death, assessed approximately up to 30 months
  Duration of response will be calculated from the date of first documentation of response per RECIST v.1.1 (complete or partial response, whichever comes first) to the date of documented PD or death. The censoring rules defined above for PFS will be used for DoR.
Clinical benefit | ≥3 months
  defined as percentage of evaluable patient with complete response, partial response or stable disease lasting ≥3 months, as defined by RECIST v1.1.
Overall survival | from the date of registration to the date of death or last contact; approximately 30 months
  calculated from the date of registration to the date of death (death event) or last contact (in this case, survival will be censored on that date).
Mid- and long-term survival | 12, 18 and 24 months
  will be the Kaplan-Meier estimates of the probability of being alive at these time points
Pharmacokinetics measures - plasma concentration | 8 days
  PK parameters will be evaluated in plasma by standard non-compartmental methods (compartmental modeling may be performed if appropriate).The dose-exposure relationships for maximum plasma concentration (Cmax) and any potential PK interaction of atezolizumab over PM01183 will be explored.
Pharmacogenetics measurements of genes implicated in the metabolism and/or transport of PM01183 | 1 day
  In order to explore factors that may help explain individual variability in the main PK parameters, the presence or absence of germline mutations or polymorphisms in genes that may be involved in the metabolism and/or transport of PM01183 will be analyzed in leukocyte DNA extracted from one blood sample (10 mL) obtained at any time during the study, but preferably just before treatment start in Cycle 1 along with the first PK sample
Pharmacogenomics measurements of predictive/prognostic markers of response and/or resistance to PM01183 and atezolizumab | 1 day
  In order to determine predictive/prognostic markers of response and/or resistance to PM01183 and atezolizumab, tumor samples available at baseline and blood samples (Day 1 of every cycle and end-of-treatment) wil be evaluated in all patients. In addition, on- treatment tumor samples from biopsy (4ht to 6ht weeks after treatment onset) wil be obtained and evaluated for patients cosenting to PGx sub- study.
Pharmacogenomics measures sub-study - tumor samples | one sample between 4th to 6th weeks after treatment onset
  For tumor biomarkers research, tumor samples will be collected on-treatment to be analyzed at the end of the study. The on-treatment biopsy will be optional, requiring specific patient consent.
  The on-treatment tumor samples will be compared to baseline tumor samples and the biomarker to analize are:
  PD-L1 and PD-L2 expression in tumor cells and in tumor-infiltrating immune cells, presence of CD8+ T cell and CD4+ T cell in stromal-tumor edge and inside the tumor parenchyma, tumor-infiltrating lymphocyte (TIL) density, expression of granzyme B, the activated transcription factor signal transducer and activator of transcription 1 (pSTAT1), Ki67, interferon gamma (IFNƔ), tumor necrosis factor alpha (TNF-α), cytotoxic T-lymphocyte-associated protein 4 (CTLA4), fractalkine, lymphocyte-activation gene 3 (LAG-3) and T-cell immunoglobulin and mucin protein 3 (TIM-3) by IHC;
  and Tumor mutational burden by DNAseq with Foundation One (or another similar validated panel).
Pharmacokinetics measures - area under the curve | 8 days
  PK parameters will be evaluated in plasma by standard non-compartmental methods (compartmental modeling may be performed if appropriate).The area under the curve (AUC) will be evaluated, and any potential PK interaction of atezolizumab over PM01183 will be explored.
Pharmacogenomics measures sub-study - blood samples | First day of each cycle (each cycle is 21 days) and at the End of Treatment visit, which is up to 37 days after the last study treatment administration
  For those patients specifically consenting, blood samples for the evaluation of biomarkers will be drawn just before treatment on Day 1 of each cycle and at EOT.
  The biomarker to analize are:
  • Plasma cytokine analysis by enzyme-linked immunosorbent assay (ELISA): IFNƔ, TNF-α, interleukins IL-1β, IL-6 and IL-18, and CXCL11 (ITAC).

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Ponce, MD, Principal Investigator — Hospital 12 de Octubre
Locations (13):
- Spain (13):
  - Hospital Virgen de la Victoria, Málaga, Andalusia
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital Universitario Da Coruña, A Coruña
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario Virgen de la Arrizaca, Murcia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza